CLINICAL TRIAL: NCT06892145
Title: Phase I Clinical Trial of CD19-targeting Chimeric Antigen Receptor T Lymphocyte (MC-1-50) for the Treatment of Refractory Adult Systemic Lupus Erythematosus(SLE)
Brief Title: Clinical Trial of CD19 Targeted CAR-T Cell in Refractory Adult SLE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB13
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus Erythematosus (SLE); Refractory
Keywords: CAR T-Cell therapy; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MC-1-50 (Experimental): Patients will be be treated with CD19 CAR- T cells
  Interventions: Biological: MC-1-50

INTERVENTIONS:
Biological: MC-1-50 — A single infusion of CD19 CAR-T cells will be administered intravenously after lymphodepletion chemotherapy

SUMMARY:
This is a single-arm, open, dose-increasing and dose-expanding phase I clinical trial to investigate the safety, tolerability and cytodynamic characteristics of MC-1-50 cell preparation, and to preliminatively observe the efficacy of MC-1-50 cell preparation in patients with refractory SLE, and to explore the applicable dose regimen for phase II clinical trials.

DETAILED DESCRIPTION:
Based on the specific CD19-targeting CAR-T developed by PrimeCARTM platform, the cell preparation time is about 3 days, which can greatly shorten the waiting time of patients, improve production efficiency and reduce production costs.At the same time, MC-1-50 products contain a high proportion of T naive cells, which can play a therapeutic role at a very low infusion dose and improve safety.

In this study, three dose groups were composed of 0.3×10^5/kg, 1×10^5/kg and 3×10^5/kg CAR-positive cells, respectively.All subjects received only one infusion of MC-1-50 cells.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or their guardian agrees to participate in this clinical trial and sign the ICF, indicating their understanding of the purpose and procedures of this clinical trial and willingness to participate in the study;
2. Age ≥ 18 years old , gender not limited;
3. Patients diagnosed with SLE according to the 2019 EULAR/ACR classification criteria,And by hydroxychloroquine, sufficient glucocorticoid (≥1mg/kg/d prednisone or equivalent amount of other hormones), to less than 2Treatment with immunosuppressants (including cyclophosphamide, motecophanate, azathioprine, methotrexate, cyclosporine, tacrolimus, sirolimus, leflunomide, etc.), and at least one approved biological agent (including titacept, Beliuzumab, etc.), with a total duration of treatment ≥3 months, still in a disease active state, or unable to tolerate conventional therapy;
4. SLEDAI-2K score ≥7 points;
5. Autoantibody test results are positive: ANA antibody positive and/or serum anti-DSDNA positive;
6. Adequate renal, hepatic, pulmonary and cardiac function defined as:

   1. Cardiac function: Echocardiography indicates left ventricular ejection fraction ≥ 50%;
   2. Renal function: serum creatinine ≤ 2.0 × ULN, or creatinine clearance rate ≥ 60ml/min (Cockcroft Gault formula);
   3. Hepatic function: ALT and AST ≤ 3.0 × ULN (may be relaxed to ≤ 3.0 × ULN in cases of combined liver infiltration);
   4. Total bilirubin ≤ 2.0 × ULN (Gilbert syndrome requires total bilirubin ≤ 3.0 × ULN);
   5. Pulmonary function: Blood oxygen saturation is ≥ 92% in non oxygen state.
7. No serious mental disorders;
8. Meet standards for apheresis or venous blood collection, and no other cell collection contraindications;
9. Women of childbearing age who have a negative blood pregnancy test and all subjects agree to use reliable and effective contraceptive methods (excluding safe period contraception) for contraception within one year after receiving MC-1-50 cell infusion from the time of signing the informed consent form. Including but not limited to: abstinence, implantable progestogen contraceptives that can inhibit ovulation; Intrauterine device (IUD); Intrauterine hormone release system; Spouse vasectomy; Compound hormone contraceptives that can inhibit ovulation (oral, vaginal, and transdermal); Progesterone contraceptives (oral or injectable) that can inhibit ovulation; When male subjects have sex with fertile women, they must agree to use barrier contraception (such as condom plus spermicidal foam/gel/film/emulsion/suppository). At the same time, participants should commit not to donate eggs (oocytes, oocytes) or sperm for assisted reproduction within one year after cell infusion.

Exclusion Criteria:

1. There were severe active central nervous system lupus that required therapeutic intervention at the time of screening;
2. Acute severe nephritis: had or was undergoing renal replacement therapy within 3 months prior to reinfusion, or had significant renal deterioration that the investigator believed was likely to cause the subject to require high doses of corticosteroids (prednisone ≥1mg/kg/ day or equivalent of other hormones), cyclophosphamide, or mycophanate during the first 3 months of the study;Clinical stable lupus nephritis that can be controlled during screening can be considered;
3. There were other lupus crises that were not controlled at the time of screening;
4. Individuals who have received CAR-T therapy or other gene modified cell therapies;
5. Combined with other autoimmune diseases requiring systemic treatment;
6. HBsAg or HBcAb positive and HBV DNA test greater than the normal range;HCV antibody positive and HCV RNA detection greater than the normal range;HIV antibody positive;Treponema pallidum antibody positive;
7. Suffered from any of the following heart diseases:

   1. New York Heart Association (NYHA) stage III or IV congestive heart failure;
   2. Within the 6 months prior to enrollment, there has been a myocardial infarction, or a coronary artery bypass grafting (CABG) or stent implantation surgery has been performed;
   3. History of ventricular arrhythmias requiring treatment or unexplained syncope (excluding cases caused by vasovagal or dehydration);
   4. History of severe non-ischemic cardiomyopathy;
8. Uncontrollable infection in the 1 weeks before enrollment;
9. History of solid organ transplantation or hematopoietic stem cell transplantation prior to screening；
10. Cerebrovascular accident or seizure occurred within 6 months prior to screening；
11. Deep vein or deep artery embolism event within the past 6 months prior to screening;
12. history of malignant neoplasms (other than tumors with no active lesion and ending treatment > 2 years ago, and adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery);
13. (attenuated) Live vaccine ≤ 4 weeks prior to screening;
14. Have participated in other clinical trials within one month or five drug half lives (whichever is shorter) before enrollment;
15. Women who are pregnant or breastfeeding, and male or female subjects who plan to have children within 1 year after receiving MC-1-50 cell infusion;
16. Other situations considered by the investigator to be unsuitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-05-04 (Estimated); Study Completion 2028-02-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 1 month
  Dose-limiting toxicity after CD19 CAR-T cell infusion
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 1 month
  The incidence of adverse events after CAR-T cell infusion was assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 5.0)

SECONDARY OUTCOMES:
Validity endpoint of MC-1-50 cells [Efficacy] | 3 months
  3M SRI-4 response rate, 6M LLDAS, DORIS response rate，SLEDAI-2K score, PGA, and BILAG-2004 change from baseline
AUCS of MC-1-50 cells [Cell dynamics] | 3 months
  AUCS is defined as the area under the curve in 28/90 days
CMAX of MC-1-50 cell preparation [Cell dynamics] | 3 months
  CMAX is defined as the highest concentration of MC-1-50 cells expanded in peripheral blood
TMAX of MC-1-50 cell preparation[Cell dynamics] | 3 months
  TMAX is defined as the time to reach the highest concentration
Pharmacodynamics of MC-1-50 cell preparation[Cell dynamics] | 3 months
  The clearance degree of CD19-positive B cells in peripheral blood was detected by flow cytometry at the visit points specified in the research protocol
Immunogenicity of pCAR-19B cells | 3 months
  The anti-CAR antibody was detected by ELISAt the visit points specified in the research protocol

OTHER OUTCOMES:
Response rate after MC-1-50 infusion [Long-term Efficacy] | 2 years
  The DORIS response rate, LLDAS maintenance rate, and SRI-4 response rate at the remaining sites after reinfusion when other drugs (including hormones, hydroxychloroquine, immunosuppressants, and biologics) were discontinued.And changes from baseline in SLEDAI-2K scores, PGA scores, BILAG-2004 scores, and serological indicators, including anti-DSDNA, anti-nuclear antibodies, and complement C3 and C4 levels
The rebuilding of the immune system | 2 years
  Proportion of B-cell subtypes at each site and their association with reduced disease activity

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital), Hefei, Anhui
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No